CLINICAL TRIAL: NCT07352306
Title: The Efficacy of Topical Diacerein Cream in Patients With Psoriasis Vulgaris
Brief Title: Topical Diacerein in Psoriasis Vulgaris
Acronym: DIA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ashraf Muhammad Helal, Teaching Assistant, Clinical Pharmacy Department, Faculty of Pharmacy, Ahram Canadian University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP 3.2.1
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis Vulgaris
Keywords: Diacerein; Psoriasis vulgaris; Topical; Interleukin-1β inhibitor; Randomized controlled trial
MeSH Terms: interventions — diacerein

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, randomized, double-blind, parallel-arm, placebo-controlled clinical trial. Participants will be randomly assigned in a 1:1 ratio to receive either topical diacerein cream or a matching placebo cream. Participants will remain in their assigned treatment arm for the duration of the study, with outcomes assessed according to the prespecified schedule. No crossover between treatment arms is planned.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to study groups using a computer-generated allocation sequence. Allocation concealment will be ensured through the use of sequentially numbered, opaque, sealed envelopes prepared by an independent individual and opened only after eligibility confirmation and informed consent.
  The investigational product and placebo will be identical in appearance and texture and prepared by qualified study personnel. Both participants and treating clinicians will remain blinded to treatment assignment for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Diacerein (Experimental): Participants assigned to this arm will receive topical diacerein cream 1% applied twice daily for a treatment period of two months.
  Interventions: Drug: Diacerein
- Placebo (Placebo Comparator): Participants assigned to this arm will receive a matching placebo topical cream applied twice daily for a treatment period of two months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerein — Topical diacerein cream 1% will be applied to affected skin areas twice daily for a treatment duration of two months.
  Other Names: Topical diacerein
  Arms: Topical Diacerein
Drug: Placebo — A matching placebo topical formulation will be applied to affected skin areas twice daily for a treatment duration of two months.
  Other Names: Matching placebo topical formulation
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of topical diacerein in adults with psoriasis vulgaris. The primary objective of the study is to compare the proportion of participants who achieve a clinically meaningful improvement in disease severity between the topical diacerein group and the placebo group.

Participants will:

Be assigned to receive topical diacerein 1% or placebo twice daily for a treatment period of 2 months.

Attend follow-up visits at Weeks 2, 4, 6, and 8. Undergo an additional evaluation one month after treatment cessation.

DETAILED DESCRIPTION:
This is a phase IV, randomized, placebo-controlled, double-blind clinical study designed to evaluate the efficacy and safety of topical diacerein in adults with psoriasis vulgaris. Participants who meet eligibility criteria will be randomized to receive either topical diacerein or matching placebo. The study treatment will be applied twice daily for two months. Participants will attend follow-up visits at Weeks 2, 4, 6, and 8, during which clinical evaluations, safety assessments, and efficacy measurements will be conducted.

The primary efficacy endpoint is the proportion of participants achieving at least a 75% improvement from baseline in the Psoriasis Area and Severity Index (PASI 75) at Week 8. Secondary endpoints may include additional PASI response thresholds, investigator global assessments, patient-reported outcomes, and safety endpoints. Safety will be monitored throughout the study through the collection of adverse events, physical examinations, and other relevant clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old of both genders.
* Patients with mild chronic plaque psoriasis body surface area (BSA < 10%) along with Psoriasis Area and Severity Index (PASI) score of < 10, and/or Dermatology Life Quality Index (DLQI) score of <10.

Exclusion Criteria:

* Documented hypersensitivity or idiosyncratic reaction to the investigational product or any excipients contained within the cream formulation.
* Intake of anti-psoriatic systemic therapy within the last 3 months, or topical treatments within the last 2 weeks.
* Patients with pustular psoriasis.
* Pregnant and breast-feeding individuals.
* Patients with psoriatic arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving PASI 75 | Week 8
  The proportion of participants who achieve at least a 75% improvement from baseline in the Psoriasis Area and Severity Index (PASI 75), comparing the topical diacerein group with the placebo group.

SECONDARY OUTCOMES:
Proportion of Participants Achieving IGA/Body-IGA Success | Week 8
  The proportion of participants achieving Investigator's Global Assessment (IGA) or Body-IGA success, defined as a score of clear or almost clear with at least a 2-grade improvement from baseline
Proportion of Participants Achieving PASI 90 | Week 8
  The percentage of participants achieving at least a 90% improvement from baseline in the Psoriasis Area and Severity Index (PASI 90).
Proportion of Participants Achieving DLQI ≤5 | Week 8
  Percentage of participants with a Dermatology Life Quality Index (DLQI) total score of ≤5.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al-Ainy Psoriasis Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data (IPD) has not yet been finalized. The availability of IPD will be determined at a later date based on ethical approvals, participant consent, data protection requirements, and institutional and sponsor policies.

REFERENCES:
- [Background] Armstrong AW, Lee K, Yee D, Woodbury M, Zundell M, Zagona-Prizio C, Yousif J, Grant C, Shields A, Chou P, Callis Duffin K, Gottlieb AB, Merola JF, Perez-Chada L. Validation of DermSat-7 for Assessing Treatment Satisfaction in Patients With Psoriasis. JAMA Dermatol. 2025 Feb 26;161(4):416-20. doi: 10.1001/jamadermatol.2024.6567. Online ahead of print. PMID 40009402
- [Background] Nael, S., M. Abbassi, and S. Farid, MSR225 Translation and Cultural Adaptation of Four EQ Bolt-Ons for the Use in the Quantitative Psychometric Investigation in Egyptian Patients With Chronic Skin Conditions. Value in Health, 2024. 27(12): p. S482.
- [Background] Napoli, G.D., Diacerein for use in treating psoriasis. 2003.
- [Background] Lebwohl MG, Kircik LH, Moore AY, Stein Gold L, Draelos ZD, Gooderham MJ, Papp KA, Bagel J, Bhatia N, Del Rosso JQ, Ferris LK, Green LJ, Hebert AA, Jones T, Kempers SE, Pariser DM, Yamauchi PS, Zirwas M, Albrecht L, Devani AR, Lomaga M, Feng A, Snyder S, Burnett P, Higham RC, Berk DR. Effect of Roflumilast Cream vs Vehicle Cream on Chronic Plaque Psoriasis: The DERMIS-1 and DERMIS-2 Randomized Clinical Trials. JAMA. 2022 Sep 20;328(11):1073-1084. doi: 10.1001/jama.2022.15632. PMID 36125472
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research Involving Human Participants. JAMA. 2025 Jan 7;333(1):71-74. doi: 10.1001/jama.2024.21972. PMID 39425955
- [Background] Wally V, Hovnanian A, Ly J, Buckova H, Brunner V, Lettner T, Ablinger M, Felder TK, Hofbauer P, Wolkersdorfer M, Lagler FB, Hitzl W, Laimer M, Kitzmuller S, Diem A, Bauer JW. Diacerein orphan drug development for epidermolysis bullosa simplex: A phase 2/3 randomized, placebo-controlled, double-blind clinical trial. J Am Acad Dermatol. 2018 May;78(5):892-901.e7. doi: 10.1016/j.jaad.2018.01.019. Epub 2018 Feb 2. PMID 29410318
- [Background] Baxi, K., et al., Diacerein in the treatment of chronic plaque psoriasis: A case report. Indian Journal of Drugs in Dermatology, 2022. 8(2): p. 79-82.
- [Background] Hu P, Wang M, Gao H, Zheng A, Li J, Mu D, Tong J. The Role of Helper T Cells in Psoriasis. Front Immunol. 2021 Dec 15;12:788940. doi: 10.3389/fimmu.2021.788940. eCollection 2021. PMID 34975883
- [Background] Elkalla N, Elhamammsy MH, Bedair NI, Elazazy O, El Kholy AA. A Promising Approach to Psoriasis Vulgaris Management with N-Acetylcysteine and Vitamin E: Targeting the Interplay of Inflammatory and Oxidative Stress. Biomedicines. 2025 May 22;13(6):1275. doi: 10.3390/biomedicines13061275. PMID 40563994
- [Background] Ramic L, Sator P. Topical treatment of psoriasis vulgaris. J Dtsch Dermatol Ges. 2023 Jun;21(6):631-642. doi: 10.1111/ddg.15042. Epub 2023 May 26. PMID 37235479
- [Background] Brunner SM, Ramspacher A, Rieser C, Leitner J, Heil H, Ablinger M, Tevini J, Wimmer M, Koller A, Pinon Hofbauer J, Felder TK, Bauer JW, Kofler B, Lang R, Wally V. Topical Diacerein Decreases Skin and Splenic CD11c+ Dendritic Cells in Psoriasis. Int J Mol Sci. 2023 Feb 21;24(5):4324. doi: 10.3390/ijms24054324. PMID 36901755